CLINICAL TRIAL: NCT01574872
Title: Double-blind, Randomized, Placebo Controlled Study Evaluating the Efficacy of Aerosal® in the Treatment of Inverse Psoriasis and Sebopsoriasis
Brief Title: Efficacy of Aerosal® in the Treatment of Inverse Psoriasis and Sebopsoriasis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Changes in the sponsorship, design and locations of the study
Sponsor: Tecno Sun SRL (Industry)
Collaborators: Centro Studi Gised (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AEROSAL1
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Inverse Psoriasis; Sebopsoriasis
Keywords: psoriasis; salt; sodium chloride
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerosal (Experimental): This arm include all patients treated with Aerosal®
  Interventions: Device: Halotherapy
- Placebo (Placebo Comparator): This arm include all patients treated with placebo
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Halotherapy — The treatment consist of 15 session of micronized iodized salt (sodium chloride) skin exposure in a chamber that reproduces the environmental characteristics of a natural salt cave. Each daily session last 30 minutes.
  Other Names: aerosal; salt; sodium chloride
  Arms: Aerosal
Device: Placebo — The treatment consist of 15 sessions in a chamber that emulates the environmental characteristics of a natural salt cave but with no salt emanation. Each daily session last 30 minutes.
  Other Names: comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of Aerosal® compared to placebo in the prognosis of inverse psoriasis or sebopsoriasis present for at least one year

ELIGIBILITY:
Inclusion Criteria:

* Inverse Psoriasis or Sebopsoriasis lasting from at one year
* At least 1% of total body surface area involvement Suspension for more than 3 months from start of the study of any systemic drugs for psoriasis, immunosuppressive treatments (cyclosporin, systemic steroids), psoralen plus ultraviolet A irradiation (PUVA) or ultraviolet B phototherapy (UVB)

Exclusion Criteria:

* Patients with acute bronchopulmonary disease, tuberculosis, severe hypertension, hyperthyroidism, cancer (chemotherapy), intoxication, heart failure
* Iodine allergy
* Women who are pregnant or planning to become pregnant during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline of PASI index equal to or greater than 50% (PASI50 +) | 3 weeks (15 sessions), 15 weeks

SECONDARY OUTCOMES:
Any change from baseline of physician's clinical judgment | 3 weeks (15 sessions), 15 weeks
  Any change from baseline of physician's clinical judgment as assessed by visual analogue scale (VAS)
Overall patient satisfaction | 3 weeks (15 sessions), 15 weeks
  Overall patient satisfaction as assessed by visual analogue scale VAS
Any change from baseline of PASI index | 3 weeks (15 sessions), 15 weeks
Number of reported adverse events | 3 weeks (15 sessions), 15 weeks
  Number of reported adverse events (AEs) during treatment period or after the end of treatment, if suspected to be related with it

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Naldi, MD, Principal Investigator — Centro Studi Gised
Locations (1):
- Fondazione S.Raffaele del Monte Tabor, Milan, Italy